CLINICAL TRIAL: NCT05011383
Title: High-dose Testosterone in Men With Metastatic Castration-resistant Prostate Cancer and ATM or CDK12 Deficiency
Brief Title: High Dose Testosterone for ATM, CDK12 or CHEK2 Altered Prostate Cancers
Acronym: VA-BAT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPLP-003-20F
Record Dates: First submitted 2021-08-11; First posted 2021-08-18 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Prostate Cancer
Keywords: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Testosterone

STUDY DESIGN:
Intervention Model Description: 3 cohort phase II study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ATM (Experimental): Patients with castration resistant prostate cancer which contains ATM alterations are treated with high dose testosterone
  Interventions: Drug: High dose testosterone
- CDK12 (Experimental): Patients with castration resistant prostate cancer which contains CDK12 alterations are treated with high dose testosterone
  Interventions: Drug: High dose testosterone
- CHEK2 (Experimental): Patients with castration resistant prostate cancer which contains CHEK2 alterations are treated with high dose testosterone
  Interventions: Drug: High dose testosterone

INTERVENTIONS:
Drug: High dose testosterone — High dose testosterone is administered subcutaneously once monthly until progression or toxicity
  Other Names: Bipolar androgen therapy

SUMMARY:
This study will determine whether the presence of DNA repair deficiency in the form of alterations in the genes ATM, CDK12 or CHEK2 predicts for a high likelihood of responding to the use of intermittent high dose testosterone. This therapy may result in responses in tumors which are genetically unstable because of DNA repair deficiency and this is a prospective study to test that hypothesis

DETAILED DESCRIPTION:
This is an unblinded, three cohort phase II study evaluating the efficacy of high dose testosterone (BAT) for patients with mCRPC and inactivating mutations in ATM, CDK12 or CHEK2. Patients will receive BAT until disease progression or intolerance, whichever occurs first. Throughout the study, safety and tolerability will be assessed by frequent recording of adverse events, vital signs and safety laboratory assessments. Progression will be evaluated with bone scan, CT of the abdomen/pelvis and PSA as per PCWG3 criteria.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form (ICF) providing agreement to adhere to the dosing schedule, report for all trial visits and authorization, use and release of health and research trial information
* Male age > 18 years
* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Ongoing gonadal androgen deprivation therapy with gonadotropin-releasing hormone (GnRH) analogues, antagonists or orchiectomy. Patients who have not had an orchiectomy must be maintained on effective GnRH analogue/antagonist therapy
* Castration resistant prostate cancer as defined by serum testosterone < 50 ng/ml and one of the following:

  * PSA level of at least 2 ng/ml that has risen on at least 2 successive occasions at least 1 week apart.
  * Evaluable disease progression by modified RECIST 1.1 (Response Evaluation Criteria in Solid Tumors)
  * Progression of metastatic bone disease on bone scan with > 2 new lesions
* Presence of metastatic disease on bone or CT scan
* Patients must have progressed on 1 next-generation AR-signaling inhibitor (e.g. abiraterone, enzalutamide, apalutamide, darolutamide, etc.).
* Asymptomatic or minimal cancer related symptoms
* Eastern Cooperative Oncology Group (ECOG) Performance Status of < 2
* Presence of inactivating mutations in ATM, CDK12 or CHEK2 as determined by a CLIA level assay for DNA sequencing.

Exclusion Criteria:

* Currently receiving active therapy for other neoplastic disorders will not be eligible.
* Histologic evidence of small cell carcinoma (morphology alone - immunohistochemical evidence of neuroendrocrine differentiation without morphologic evidence is not exclusionary)
* Known parenchymal brain metastasis
* Liver metastases
* Active or symptomatic viral hepatitis or chronic liver disease AST or ALT > 2.5 x ULN or total bilirubin > ULN (unless Gilbert's syndrome is the etiology of hyperbilirubinemia).
* Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) Class II-IV heart disease or cardiac ejection fraction measurement of <35 % at baseline
* Patients with pain attributable to their prostate cancer and requiring the use of opioids.
* Tumor causing urinary outlet obstruction that requires catheterization for voiding. Patients that require catheterization to void secondary to benign strictures or other non-cancer causes will be permitted to enroll.
* Presence of dementia, psychiatric illness, and/or social situations limiting compliance with study requirements or understanding and/or giving of informed consent.
* Any condition(s), medical or otherwise, which, in the opinion of the investigators, would jeopardize either the patient or the integrity of the data obtained.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer only develops in males
Enrollment: 51 (Estimated)
Dates: Start 2021-08-31 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
PSA response | 12 weeks
  PSA response as measured by a 50% decline from baseline maintained for 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert B. Montgomery, MD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (17):
- United States (17):
  - Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - Orlando VA Medical Center, Orlando, FL, Orlando, Florida
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Robley Rex VA Medical Center, Louisville, KY, Louisville, Kentucky
  - Kansas City VA Medical Center, Kansas City, MO, Kansas City, Missouri
  - St. Louis VA Medical Center John Cochran Division, St. Louis, MO, St Louis, Missouri
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - Salisbury W.G. (Bill) Hefner VA Medical Center, Salisbury, NC, Salisbury, North Carolina
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina
  - Memphis VA Medical Center, Memphis, TN, Memphis, Tennessee
  - Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington
  - William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No